CLINICAL TRIAL: NCT04403633
Title: Improving Patient-Centered Care in Pediatric Acute Kidney Injury (Change Peds AKI)
Brief Title: A Study of Facilitators and Barriers to Improve Acute Kidney Injury in Children Through Mobile Health Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00104197; 1R38HL143612-01 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury
Keywords: AKI; Pediatric AKI; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving Educational Tool (Experimental): Patients in this arm will receive the educational tool after the pretest in addition to usual care.
  Interventions: Other: mobile health educational tool
- Receiving Usual Care (No Intervention): Patients in this arm will receive usual care after the pretest.

INTERVENTIONS:
Other: mobile health educational tool — Interactive educational tool delivered on iPad
  Arms: Receiving Educational Tool

SUMMARY:
The purpose of this study is to improve patient-centered care for acute kidney injury (AKI) in order to decrease the adverse health outcomes associated with this common condition.

DETAILED DESCRIPTION:
There is a need to provide better patient-centered care for acute kidney injury (AKI) in order to improve the adverse health outcomes associated with this common condition. This project involves thorough evaluation of patient and provider feedback on barriers and facilitators to pediatric AKI self-management in order to develop patient-centered pediatric AKI interventions. This will be done through interviews with families of patients diagnosed with AKI and providers who take care of these patients followed by integration of the results into modification of an existing educational tool previously used in adult patients. The study will take place in three parts with the first involving interviews, the second involving tool modification and usability testing, and the third involving pilot testing of the tool's impact.

ELIGIBILITY:
Inclusion Criteria:

* age 1 to 18 years
* patients with diagnosis of AKI while hospitalized

Exclusion Criteria:

* legal blindness of deafness
* cognitive impairment that limits ability to consent
* non-English speaking
* patient age greater than age 18 years, 11 months

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) Knowledge Assessment score | Baseline, 1 month
  AKI Knowledge Assessment administered as pre-test prior to intervention and post-test one month after intervention. This assessment is scored with minimum value of 0% and maximum value of 100%. A higher score is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa J Diamantidis, MD, Principal Investigator — Duke University; Rasheed Gbadegesin, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No